CLINICAL TRIAL: NCT02389829
Title: Hydromorphone Versus Prochlorperazine + Diphenhydramine for Treatment of Acute Migraine. A Randomized, Emergency Department Based, Comparative Efficacy Study
Brief Title: Hydromorphone Versus Prochlorperazine + Diphenhydramine for Acute Migraine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Benjamin W. Friedman, MD, Associate Professor, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014-4325
Record Dates: First submitted 2015-03-10; First posted 2015-03-17 (Estimated); Results first posted 2018-06-06 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Hydromorphone; Prochlorperazine; Diphenhydramine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hydromorphone (Active Comparator): Hydromorphone 1mg, administered as intravenous drip over 5 minutes. Patients can receive second 1mg dose at 1 hour.
  Interventions: Drug: Hydromorphone
- Prochlorperazine (Active Comparator): Prochlorperazine 10mg, administered as intravenous drip over 5 minutes. Diphenhydramine 25mg co-administered.
  Patients can receive second 10mg dose at 1 hour.
  Interventions: Drug: Prochlorperazine; Drug: Diphenhydramine

INTERVENTIONS:
Drug: Hydromorphone
  Other Names: Dilaudid
  Arms: Hydromorphone
Drug: Prochlorperazine
  Other Names: Compazine
  Arms: Prochlorperazine
Drug: Diphenhydramine
  Other Names: Benadryl
  Arms: Prochlorperazine

SUMMARY:
Opioids are commonly used to treat migraine in North American Emergency Departments. We are comparing efficacy and adverse events of hydromorphone, an opioid, to that of prochlorperazine, a dopamine antagonist with known efficacy in migraine. Prochlorperazine will be combined with diphenhydramine to prevent adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Migraine headache (International Classification of Headache Disorders 3B criteria)

Exclusion Criteria:

* Brain imaging ordered
* Fever
* Objective neurological findings
* Pregnancy/ breast feeding
* Allergy/ contraindication to investigational medication
* History of addiction to opioids, use of methadone, any use of opioids previous 30 days

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2015-03; Primary Completion 2016-06 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin W Friedman, MD, MS, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center--Einstein, The Bronx, New York, United States

REFERENCES:
- [Derived] Cohen F, Friedman BW. A randomized study of IV prochlorperazine plus diphenhydramine versus IV hydromorphone for migraine-associated symptoms: A post hoc analysis. Headache. 2021 Sep;61(8):1227-1233. doi: 10.1111/head.14185. Epub 2021 Aug 7. PMID 34363617
- [Derived] Friedman BW, Irizarry E, Solorzano C, Latev A, Rosa K, Zias E, Vinson DR, Bijur PE, Gallagher EJ. Randomized study of IV prochlorperazine plus diphenhydramine vs IV hydromorphone for migraine. Neurology. 2017 Nov 14;89(20):2075-2082. doi: 10.1212/WNL.0000000000004642. Epub 2017 Oct 18. PMID 29046364

RESULTS

PARTICIPANT FLOW:
Groups:
- Hydromorphone: Hydromorphone 1mg, administered as intravenous drip over 5 minutes. Patients can receive second 1mg dose at 1 hour.
  Hydromorphone
- Prochlorperazine: Prochlorperazine 10mg, administered as intravenous drip over 5 minutes. Diphenhydramine 25mg co-administered.
  Patients can receive second 10mg dose at 1 hour.
  Prochlorperazine
  Diphenhydramine
Period: Overall Study
Arm/Group | Hydromorphone | Prochlorperazine
Started | 64 | 63
Completed | 64 | 62
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydromorphone | Prochlorperazine | Total
Number analyzed (Participants) | 64 | 63 | 127
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (11) | 32 (9) | 34 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 50 | 106
  Male | 8 | 13 | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 64 | 63 | 127
Duration of headache Prior to Study [Median (Inter-Quartile Range); unit: Hours] | 48 [24 to 96] | 72 [24 to 96] | 48 [24 to 96]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Sustained Headache Relief Assessed by Self-evaluation
Description: Sustained headache relief is defined as achieving a headache level of "mild" or "none" within two hours and maintaining a level of "mild" or "none" for 48 hours, without use of addition medication. Patient self-evaluated pain level is solicited every half hour for two hours in the Emergency Department and then by telephone 48 hours after medication administration.
Time Frame: up to 2 hours in Emergency Department, 48 hours after discharge from Emergency Department
Measure: Count of Participants; unit: Participants
Arm/Group | Hydromorphone | Prochlorperazine
Number analyzed (Participants) | 64 | 63
Participants | 20 | 37

2. Secondary Outcome: Number of Participants Needing Rescue Medication as Assessed by Questionnaire
Description: Data collected by telephone. Patients were asked if they needed additional medication after discharge in order to reduce level of pain. This additional medication is considered rescue medication.
Time Frame: 48 hours after discharge from Emergency Department
Measure: Count of Participants; unit: Participants
Arm/Group | Hydromorphone | Prochlorperazine
Number analyzed (Participants) | 64 | 63
Participants | 23 | 4

3. Secondary Outcome: Number of Participants Who Achieved Short Term Headache Relief, Assessed by Telphone Questionnaire
Description: Participants were asked to make evaluation of pain status since discharge. Those achieving headache level "mild" or "none" for 1 hour are considered to achieve short term headache relief.
Time Frame: 48 hours after discharge from Emergency Department
Measure: Count of Participants; unit: Participants
Arm/Group | Hydromorphone | Prochlorperazine
Number analyzed (Participants) | 64 | 62
Participants | 33 | 53

4. Secondary Outcome: Number of Participants Who Achieved Short Term Headache Freedom; Assessed by Telephone Questionnaire
Description: Participants were asked to evaluate pain status since discharge. Participants who achieved total headache freedom for at least 1 hour are considered to achieve short term headache relief.
Time Frame: 48 hours after discharge from Emergency Department
Measure: Count of Participants; unit: Participants
Arm/Group | Hydromorphone | Prochlorperazine
Number analyzed (Participants) | 64 | 63
Participants | 16 | 29

ADVERSE EVENTS:
Time Frame: Adverse events were assessed by patient-initiated reports. In several cases, the explicit adverse event name/description was not documented. These events were grouped into the category called "other". Adverse events assessed over 48 hours post-treatment.
Arm/Group | Hydromorphone | Prochlorperazine
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/63
Other Adverse Events (participants affected / at risk) | 13/64 | 7/63
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydromorphone (N=64) | Prochlorperazine (N=63)
Dizzy (Nervous system disorders) | 9 (9) | 0 (0)
Restlessness (General disorders) | 0 (0) | 3 (3)
Other (General disorders) | 4 (4) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes